CLINICAL TRIAL: NCT05668533
Title: Comparing Postoperative Analgesic Efficiency of Intrscalene Block Versus Pericapsular Nerve Group Block for Arthroscopic Shoulder Surgery: A Randomized Controlled Clinical Trial
Brief Title: Intrscalene Block Versus Pericapsular Nerve Group Block for Arthroscopic Shoulder Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, rehab zayed, Ass. Professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0305847
Record Dates: First submitted 2022-12-10; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Rotator Cuff; Bankert Repair

STUDY DESIGN:
Intervention Model Description: 1. Interscalene group: Patients received ipsilateral ultrasound-guided interscalene nerve after induction of general anesthesia using bupivacaine 0.25% (0.5 mL/kg).
  2. PENG Block: Patients received ultrasound-guided PENG block after induction of general anesthesia using bupivacaine 0.25% (0.5 mL/kg).
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Interscalene group (Active Comparator): Patients received ipsilateral ultrasound-guided interscalene nerve after induction of general anesthesia using bupivacaine 0.25% (0.5 mL/kg).
  Interventions: Diagnostic Test: Interscalene versus PENG Block
- 2. PENG Block (Active Comparator): Patients received ultrasound-guided PENG block after induction of general anesthesia using bupivacaine 0.25% (0.5 mL/kg).
  Interventions: Diagnostic Test: Interscalene versus PENG Block

INTERVENTIONS:
Diagnostic Test: Interscalene versus PENG Block — 1. Interscalene group: Patients received ipsilateral ultrasound-guided interscalene nerve after induction of general anesthesia using bupivacaine 0.25% (0.5 mL/kg).
  2. PENG Block: Patients received ultrasound-guided PENG block after induction of general anesthesia using bupivacaine 0.25% (0.5 mL/kg).

SUMMARY:
Early postoperative pain after arthroscopic shoulder surgery is a major problem for patients and orthopedic surgeons. Adequate pain control is vital for all aspects of patient recovery; including mental state, nutrition, cost of care period, rehabilitation, patient satisfaction, and overall post-surgery outcomes. (1) Single analgesic regimens are not always effective in controlling moderate to severe postoperative pain. Therefore, multimodal pain management is preferred and is currently recommended for early postoperative pain control.(2) Regional techniques form an integral part of multimodal analgesia of most of the enhanced recovery protocols and aid in minimizing the requirements of opioids to control acute postoperative pain which results in better, faster recovery and better satisfaction. Also, it is well known that sufficient management of acute pain is essential to prevent its transition to chronic pain.(3) The use of ultrasound guidance and its incorporation into the practice of regional anesthesia has dramatically improved the safety and success of perioperative care.(4) Ultrasound guided regional anesthesia is preferred in shoulder surgery as an effective way to provide anesthesia and postoperative analgesia. To ensure adequate postoperative pain control, nerve supply to the synovium, capsule, joint surfaces, ligaments, periosteum and shoulder muscles must be blocked.

Interscalene brachial plexus (ISB) block is considered the analgesic technique of choice for shoulder surgery. However, the hemi-diaphragmatic paresis that may occur after the block has led to the search for an alternative to the ISB block. (5) Pericapsular nerve group block (PENG) is a new block that provides a pericapsular distribution with local anesthetic infiltration around the glenohumeral joint and provides analgesia by reaching the sensory nerve branches of the glenohumeral joint. The block of this area did not cause motor block or pulmonary complications, nor result in muscle laxity, blocking only the shoulder and the upper third of the humerus. It was demonstrated that the PENG block may be safely applied for both partial anesthesia and analgesia.(6)

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status class I - II
* patient who will be scheduled for an elective unilateral arthroscopic shoulder surgery

Exclusion Criteria:

* Patients with respiratory disease, renal or hepatic insufficiency,
* infection of the skin in the puncture area,
* coagulopathy,
* allergy against any of the drugs to be used (bupivacaine),
* neuromuscular disease,
* obesity (body mass index, BMI >30),
* previous analgesic medication, chronic pain, and previously known neurological pathologies or central nervous system disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | 24 hours postoperative
  visual analogue scale to assess the analgesic efficacy of ultrasound-guided intrscalene block versus PENG Block

CONTACTS AND LOCATIONS:
Locations (1):
- Rehab A. Abd El-Aziz, Alexandria, Egypt